CLINICAL TRIAL: NCT06633744
Title: Laparoscopic Versus Open Appendectomy Plus Peritoneal Lavage for Acute Complicated Appendicitis Patients With Diffuse Peritonitis: A Single-center Retrospective Study
Brief Title: Laparoscopic Versus Open Appendectomy Plus Peritoneal Lavage for Acute Complicated Appendicitis Patients With Diffuse Peritonitis
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-07
Record Dates: First submitted 2024-10-06; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Acute Complicated Appendicitis With Diffuse Peritonitis
Keywords: Acute appendicitis, Laparoscopic appendectomy, Open appendectomy Peritoneal lavage, Diffuse peritonitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aim to evaluate the efficacy and safety of laparoscopic versus open appendectomy in the treatment of acute complicated appendicitis with diffuse peritonitis.

DETAILED DESCRIPTION:
Appendicitis is defined as inflammation of the vermiform appendix and worldwide is the most common reason for emergency abdominal surgery. Globally, the annual incidence is 96.5 to 100 cases per 100 000 adult population. For acute uncomplicated appendicitis, antibiotic therapy has emerged as the primary treatment, often allowing patients to avoid surgery. However, the management of acute complicated appendicitis requires careful consideration of various treatment options.

Complicated appendicitis, characterized by peri-appendiceal phlegmon or abscess formation, presents additional challenges and often requires a more comprehensive treatment approach. Management strategies have evolved to incorporate both conservative and surgical treatments, tailored to the patient's condition. However, for Acute complicated appendicitis with diffuse peritonitis, surgery is the only option. Acute complicated appendicitis with diffuse peritonitis is a severe abdominal emergency that often requires prompt surgical intervention. Traditionally, open appendectomy has been the standard approach. In recent years, laparoscopic appendectomy has gained popularity due to its minimally invasive nature and potential for faster recovery. Despite this, the optimal surgical approach for complicated appendicitis with diffuse peritonitis remains debated, particularly regarding the risk of postoperative complications and recovery outcomes. The primary aim of this study is to compare the efficacy and safety of laparoscopic versus open appendectomy in such cases, focusing on postoperative complications, hospital stay, and other factors influencing surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 or older;

Patients with diffuse peritonitis caused by a perforated appendix confirmed intraoperatively;

Patients who underwent emergency appendectomy with peritoneal lavage;

Patients who had postoperative pathological confirmation of acute appendicitis.

-

Exclusion Criteria:

Patients younger than 18 years;

Patients have a history of prior malignancies;

Patients with incomplete clinical or pathological records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute complicated appendicitis patients with diffuse peritonitis who met the criteria.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy and safety of laparoscopic versus open appendectomy in the treatment of acute complicated appendicitis with diffuse peritonitis | January 01, 2025 to December 31, 2025.
  This involved analyzing the correlation between the surgical approach and the incidence of postoperative complications, particularly surgical site infections (SSI).

IPD SHARING:
Plan to Share IPD: No